CLINICAL TRIAL: NCT03848949
Title: Prospective Randomized-controlled Trial of an Orthotic Designed to Equalize Leg Lengths for Patients With Injuries Managed in Walking Boots
Brief Title: Study of an Orthotic Designed to Equalize Leg Lengths for Patients With Injuries Managed in Walking Boots
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Kamran S Hamid, MD, Orthopaedic Foot and Ankle Surgeon, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ORA: 18012208-IRB02
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Results first posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Joint Pain; Trouble Balancing
MeSH Terms: conditions — Arthralgia

STUDY DESIGN:
Intervention Model Description: Subjects are randomly assigned to two groups using a blocked randomization schedule.
  Subjects assigned to the control group receive the standard treatment for their condition, which must be at least 2 weeks of weight bearing as tolerated in a controlled ankle movement boot in order for them to meet inclusion criteria.
  Subjects assigned to the experimental group receive the orthotic for use on the contralateral limb, which is the only alteration to their treatment of at least 2 weeks of weight bearing as tolerated in a controlled ankle movement boot (required to meet inclusion criteria).
Masking Description: Both patients and surgeons are aware whether they are being assigned to the control group or the experimental group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Orthotic Group (Experimental): Subjects enrolled in the orthotic group receive the orthotic (Evenup) meant to increase the effective leg length of the uninjured limb.
  Interventions: Device: Evenup
- Control (No Intervention): Subjects enrolled in the control group receive the standard treatment associated with their injury (no orthotic)

INTERVENTIONS:
Device: Evenup — Orthotic which increases effective leg length.
  Arms: Orthotic Group

SUMMARY:
Patients who undergo foot and ankle surgery are often made weight-bearing as tolerated (WBAT) in a controlled ankle movement (CAM) boot during their recovery and rehabilitation process. However, some patients may experience pain and discomfort while wearing the CAM boot. A possible cause for this pain is that the boot elevates the injured foot higher than the other foot in the normal shoe. This uneven walking plane can lead to an abnormal gait or walking pattern, and may potentially lead to pain. Our goal is the investigate if using a leg-length-evening orthotic can improve balance and/or decrease the development of pain in the legs and spine for patients who are WBAT in a CAM boot.

DETAILED DESCRIPTION:
Patients with foot and ankle injuries are often made weight-bearing as tolerated (WBAT) in a controlled ankle movement (CAM) boot at some point during their recovery and rehabilitation period. While WBAT in a CAM boot, patients often experience an asymmetric gait associated with the effective leg length discrepancy between the booted extremity (longer) and the contralateral extremity with a regular shoe (shorter). This asymmetry may cause balance problems or place strain on the patient's joints resulting in back, knee, and hip pain.

An orthotic has been designed that is added to the outside of a regular shoe in order to eliminate the effective leg length discrepancy between the booted extremity and the contralateral limb. Although this specific orthotic has not been studied, some proof of concept lies in studies that show that back pain can be managed with foot orthotics. The purpose of this study is to determine if using the leg-length-evening orthotic can improve balance and/or decrease the development of pain in the lower extremities and spine for patients who are WBAT in a CAM boot.

ELIGIBILITY:
Inclusion Criteria:

* must be weight bearing as tolerated and treated for at least 2 weeks in a controlled ankle movement boot.

Exclusion Criteria:

* unwilling to participate
* being treated for an Achilles tendon rupture (and therefore being treated in a controlled ankle boot with heel lifts)
* member of a special population

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kamran S Hamid, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] White R, Schuren J, Wardlaw D, Diamandopoulos Z, Anderson R. Biomechanical assessment of gait in below-knee walking casts. Prosthet Orthot Int. 1999 Aug;23(2):142-51. doi: 10.3109/03093649909071626. PMID 10493142
- [Background] Ferrari R. Effect of customized foot orthotics in addition to usual care for the management of chronic low back pain following work-related low back injury. J Manipulative Physiol Ther. 2013 Jul-Aug;36(6):359-63. doi: 10.1016/j.jmpt.2013.06.002. Epub 2013 Jul 3. PMID 23830710
- [Background] Cambron JA, Dexheimer JM, Duarte M, Freels S. Shoe Orthotics for the Treatment of Chronic Low Back Pain: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2017 Sep;98(9):1752-1762. doi: 10.1016/j.apmr.2017.03.028. Epub 2017 Apr 30. PMID 28465224
- [Background] Ferrari R. Responsiveness of the short-form 36 and oswestry disability questionnaire in chronic nonspecific low back and lower limb pain treated with customized foot orthotics. J Manipulative Physiol Ther. 2007 Jul-Aug;30(6):456-8. doi: 10.1016/j.jmpt.2007.03.016. PMID 17693336

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment continued until the study met protocol requirement.
Groups:
- Intervention Group: Patients who received the orthotic device
- Control Group: Patients who did not receive the orthotic device.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 54 | 53
Completed | 49 | 46
Not Completed | 5 | 7
Not completed — Lost to Follow-up | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Patients who received the orthotic device.
- Control: Patients who did not receive the orthotic device.
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 49 | 46 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (2.5) | 48.8 (2.33) | 47.9 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 28 | 60
  Male | 17 | 18 | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 49 | 46 | 95
Condition: malleolar fracture, foot fracture, ankle fracture, tibiotalar arthritis etc. [Count of Participants; unit: Participants]
  Malleolar fracture | 9 | 10 | 19
  Foot fracture | 9 | 8 | 17
  Ankle sprain | 6 | 8 | 14
  Tibiotalar arthritis | 8 | 1 | 9
  Posterior tibial tendon dysfunction | 3 | 4 | 7
  Acute Achilles tendon rupture | 0 | 4 | 4
  Hindfoot arthritis | 2 | 1 | 3
  Midfoot arthritis | 1 | 2 | 3
  Peroneal pathology | 2 | 1 | 3
  Ankle Impingement | 2 | 1 | 3
  Ankle instability | 2 | 0 | 2
  Foot sprain | 0 | 2 | 2
  Other | 4 | 4 | 8
  Plantar fasciitis | 1 | 0 | 1
Condition is tibiotalar or above [Count of Participants; unit: Participants]
  Condition at or proximal to tibiotalar joint | 28 | 26 | 54
  Condition predominantly below or distal to tibiotalar joint | 21 | 20 | 41
Postoperative versus nonoperative management [Count of Participants; unit: Participants]
  Postoperative | 17 | 19 | 36
  Nonoperative | 32 | 27 | 59

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Balance
Description: Patient reported assessment of their balance while wearing the controlled ankle movement boot on a scale of 1 - 10 (higher values indicate better balance).
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Orthotic Group | Control
Number analyzed (Participants) | 49 | 46
units on a scale | 3.0 (1.7) | 2.1 (1.7)

2. Primary Outcome: Patient Reported Pain
Description: Patient reported assessment of joint pain while wearing the controlled ankle movement boot on scales of 1 - 10 (higher values indicate more pain).
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Orthotic Group | Control
Number analyzed (Participants) | 49 | 46
score on a scale | 4.9 (5.6) | 3.9 (5.1)

ADVERSE EVENTS:
Time Frame: Adverse events were collected two weeks after consent/baseline.
Arm/Group | Orthotic Group | Control
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/46
Other Adverse Events (participants affected / at risk) | 0/49 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/49/NCT03848949/Prot_SAP_ICF_002.pdf